CLINICAL TRIAL: NCT02246166
Title: A Double-Blind, Randomised, Placebo-Controlled, Parallelgroup, Single-Dose Study to Evaluate Effect of Paracetamol, Pseudoephedrine Hydrochloride, Dextromethorphan Hydrobromide and Chlorpheniramine Maleate Tablets Compared to Placebo in Subjects Suffering From the Common Cold or Influenza Over a 4 Hour Period
Brief Title: The Effect of Paracetamol, Pseudoephedrine Hydrochloride, Dextromethorphan Hydrobromide and Chlorpheniramine Maleate Tablets Compared to Placebo in Subjects Suffering From the Common Cold or Influenza.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Sino-American Tianjin Smith Kline & French Laboratories Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202271; RH02565 (Other: GSK)
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-05

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test tablet (Experimental): Tablet containing Paracetamol, Pseudoephedrine Hydrochloride, Dextromethorphan Hydrobromide and Chlorpheniramine Maleate Tablets (II) (Paracetamol 500mg, pseudoephedrine 30mg, chlorpheniramine 2mg and dextromethorphan 15mg).
  Interventions: Drug: Test tablet
- Placebo (Placebo Comparator): Matching placebo tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Test tablet — The active tablet will be administered orally. Product administration will occur within 30mins of the baseline assessment of symptom severity
  Arms: Test tablet
Other: Placebo — The placebo tablet will be administered orally. Product administration will occur within 30mins of the baseline assessment of symptom severity
  Arms: Placebo

SUMMARY:
This phase IV multi-centre, randomised, double-blind, placebo-controlled, parallel-group, single-dose study will assess the efficacy and tolerability of the active tablets versus placebo in participants suffering from cold and influenza. Eligible participants will be randomly assigned to one of 2 treatment groups (active or placebo tablets) and enter a four-hour (hr) treatment phase. Each participant will be administered only once during each study period. Participants will use a questionnaire to record the symptom severity scores as described, as well as time.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years and less than 65 years
* Good general and mental health in the opinion of the investigator
* Participants diagnosed with a common cold or flu and must have the following symptoms of at least "moderate" in intensity (≥ 2) at the screening visit (baseline), with a minimum total symptom score of 6:

  (i) At least one of pain symptoms: sore throat, headache, or extremities pain (ii) Mandatory: Nasal congestion (iii) At least one of catarrh symptoms: runny nose or sneezing
* Onset of first symptoms of cold must have occurred within 48 hours of screening.

Exclusion Criteria:

* Pregnant or breast feeding women
* History of seasonal or perennial allergic rhinitis or acute, sub-chronic, or chronic cough due to any condition other than a common cold or flu, as determined by the investigator
* Concurrent illness or medical history that is contraindicated or cautioned about in the drug label
* Anatomical factors causing nasal congestion
* Fever with body temperature >38.5°C at baseline
* Have used any medication or herbal remedies to treat cold prior to screening (antibiotics in the last 7 days, antihistamines in the last 72 hours, analgesics or antipyretics in the last 24 hours, decongestant in the last 12 hours, antitussive, medicated lozenge or throat spray in the last 8 hours)
* Any medication that has potential drug-drug interactions with study medications
* Known or suspected intolerance or hypersensitivity to the study materials
* Have a positive drug urine test or recent history (within the last 2 years) of alcohol or other substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited at 2 clinical sites in China
Period: Overall Study
Arm/Group | Test Tablet | Placebo
Started | 26 | 27
Completed | 25 | 27
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall participants in the test arm were 25 as 1 participant data was not included in the baseline measure as he did not completed the study (Due to protocol deviation).
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Tablet | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (11.97) | 38.5 (11.06) | 38.2 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Symptom Severity Assessment at 15 Minutes
Description: Symptom severity assessment was determined by Total Sum Score (TSS), TSS ranged from 0 to 21 with less severity score at the given time point represented a better outcome measure.
  TSS was calculated as the sum of the non missing scores (all on a 0-3 scale measuring worsening or severity) of the following common cold symptoms: sore throat, headache, extremities pain, nasal congestion, runny nose, sneezing, and cough post treatment administration.
  Participants self assessed symptoms severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at 15 minutes post product use.
Time Frame: 15 minutes
Population: The primary population for assessment of efficacy was the intent to treat (ITT) population. The ITT population was defined as all participants who were randomized and received at least one dose of treatment during the study and provide at least one post baseline assessment of efficacy.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Observed value | 10.66 (0.309) | 10.64 (0.304)
  Change from baseline | -1.11 (0.309) | -1.13 (0.304)
Statistical Analysis 1: Comparison: Test Tablet vs Placebo; Test type: Superiority or Other; p = 0.9473, ANCOVA; From ANCOVA model with factors for treatment group and study site and baseline TSS score as a covariate; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.77 to 0.83] — Difference is first named treatment minus the second named treatment such that a negative difference favors the first named treatment

2. Primary Outcome: Symptom Severity Assessment at 30 Minutes
Description: Symptom severity assessment was determined by TSS, TSS ranged from 0 to 21 with less severity score at the given time point represented a better outcome measure.
  TSS was calculated as the sum of the non missing scores (all on a 0-3 scale measuring worsening or severity) of the following common cold symptoms: sore throat, headache, extremities pain, nasal congestion, runny nose, sneezing, and cough post treatment administration.
  Participants self assessed symptoms severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at 30 minutes post product use.
Time Frame: 30 minutes
Population: The primary population for assessment of efficacy was the intent to treat (ITT) population. The intent-to-treat (ITT) population was defined as all participants who were randomized and received at least one dose of treatment during the study and provide at least one post baseline assessment of efficacy.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Observed value | 9.55 (0.402) | 9.74 (0.396)
  Change from baseline | -2.22 (0.402) | -2.03 (0.396)
Statistical Analysis 1: Comparison: Test Tablet vs Placebo; Test type: Superiority or Other; p = 0.7210, ANCOVA; From ANCOVA model with factors for treatment group and study site and baseline TSS score as a covariate; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-1.23 to 0.86] — Difference is first named treatment minus the second named treatment such that a negative difference favors the first named treatme

3. Primary Outcome: Symptom Severity Assessment at 1 Hour
Description: Symptom severity assessment was determined by TSS, TSS ranged from 0 to 21 with less severity score at the given time point represented a better outcome measure.
  TSS was calculated as the sum of the non missing scores (all on a 0-3 scale measuring worsening or severity) of the following common cold symptoms: sore throat, headache, extremities pain, nasal congestion, runny nose, sneezing, and cough post treatment administration.
  Participants self assessed symptoms severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at 1hour post product use.
Time Frame: 1 hour
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Observed value | 8.73 (0.495) | 8.52 (0.487)
  Change from baseline | -3.04 (0.495) | -3.25 (0.487)
Statistical Analysis 1: Comparison: Test Tablet vs Placebo; Test type: Superiority or Other; p = 0.7445, ANCOVA; From ANCOVA model with factors for treatment group and study site and baseline TSS score as a covariate; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-1.07 to 1.49]

4. Primary Outcome: Symptom Severity Assessment at 2 Hours
Description: Symptom severity assessment was determined by TSS, TSS ranged from 0 to 21 with less severity score at the given time point represented a better outcome measure.
  TSS was calculated as the sum of the non missing scores (all on a 0-3 scale measuring worsening or severity) of the following common cold symptoms: sore throat, headache, extremities pain, nasal congestion, runny nose, sneezing, and cough post treatment administration.
  Participants self assessed symptoms severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at 2 hours post product use.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Observed value | 7.54 (0.596) | 7.31 (0.587)
  Change from baseline | -4.23 (0.596) | -4.46 (0.587)
Statistical Analysis 1: Comparison: Test Tablet vs Placebo; Test type: Superiority or Other; p = 0.7662, ANCOVA; From ANCOVA model with factors for treatment group and study site and baseline TSS score as a covariate; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-1.32 to 1.78]

5. Primary Outcome: Symptom Severity Assessment at 3 Hours
Description: Symptom severity assessment was determined by TSS, TSS ranged from 0 to 21 with less severity score at the given time point represented a better outcome measure.
  TSS was calculated as the sum of the non missing scores (all on a 0-3 scale measuring worsening or severity) of the following common cold symptoms: sore throat, headache, extremities pain, nasal congestion, runny nose, sneezing, and cough post treatment administration.
  Participants self assessed symptoms severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at 3 hours post product use.
Time Frame: 3 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Observed value | 6.80 (0.669) | 6.25 (0.659)
  Change from baseline | -4.97 (0.669) | -5.52 (0.659)
Statistical Analysis 1: Comparison: Test Tablet vs Placebo; Test type: Superiority or Other; p = 0.5208, ANCOVA; From ANCOVA model with factors for treatment group and study site and baseline TSS score as a covariate; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-1.18 to 2.29] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Symptom Severity Assessment at 4 Hours
Description: Symptom severity assessment was determined by TSS, TSS ranged from 0 to 21 with less severity score at the given time point represented a better outcome measure.
  TSS was calculated as the sum of the non missing scores (all on a 0-3 scale measuring worsening or severity) of the following common cold symptoms: sore throat, headache, extremities pain, nasal congestion, runny nose, sneezing, and cough post treatment administration.
  Participants self assessed symptoms severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at 4 hours post product use.
Time Frame: 4 hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Observed value | 5.94 (0.702) | 5.82 (0.692)
  Change from baseline | -5.83 (0.702) | -5.95 (0.692)
Statistical Analysis 1: Comparison: Test Tablet vs Placebo; Test type: Superiority or Other; p = 0.8993, ANCOVA; From ANCOVA model with factors for treatment group and study site and baseline TSS score as a covariate; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-1.71 to 1.94] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Global Assessment of Treatment
Description: After completing the 4 hours symptom severity assessments, participants evaluated their treatment response on a 5-point scale by answering the question: "How well did the test medication control your symptoms?" (0-ineffective, 1-poor, 2-fair, 3-good, or 4-excellent).
Time Frame: 4 hours
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Participants
  Ineffective (0) | 1 | 2
  Poor (1) | 1 | 3
  Fair (2) | 9 | 3
  Good (3) | 10 | 17
  Excellent (4) | 4 | 2

8. Secondary Outcome: Sore Throat Severity Assessment
Description: Participants self-assessed sore throat severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at baseline and at 15, 30, 60, 120,180 and 240 minutes post product administration. All sore throat severity assessment values were recorded in questionnaire and tabulated. A reduction in severity score from baseline represented a better outcome measure.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Change from baseline in 15 minutes | -0.12 (0.076) | -0.28 (0.073)
  Change from baseline in 30 minutes | -0.21 (0.082) | -0.29 (0.080)
  Change from baseline in 60 minutes | -0.27 (0.099) | -0.29 (0.096)
  Change from baseline in 120 minutes | -0.33 (0.124) | -0.49 (0.120)
  Change from baseline in 180 minutes | -0.33 (0.132) | -0.53 (0.128)
  Change from baseline in 240 minutes | -0.46 (0.137) | -0.71 (0.133)

9. Secondary Outcome: Headache Severity Assessment
Description: Participants self-assessed headache severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at baseline and at 15, 30, 60, 120,180 and 240 minutes post product administration. All headache severity assessment values were recorded in questionnaire and tabulated. A reduction in severity score from baseline represented a better outcome measure.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Change from baseline in 15 minutes | -0.17 (0.094) | -0.14 (0.090)
  Change from baseline in 30 minutes | -0.31 (0.113) | -0.16 (0.108)
  Change from baseline in 60 minutes | -0.47 (0.130) | -0.51 (0.123)
  Change from baseline in 120 minutes | -0.72 (0.123) | -0.71 (0.117)
  Change from baseline in 180 minutes | -0.89 (0.130) | -0.88 (0.123)
  Change from baseline in 240 minutes | -0.99 (0.125) | -0.96 (0.118)

10. Secondary Outcome: Extremities Pain Severity Assessment
Description: Participants self-assessed extremities pain severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at baseline and at 15, 30, 60, 120,180 and 240 minutes post product administration. All extremities pain severity assessment values were recorded in a questionnaire and tabulated. A reduction in severity score from baseline represented a better outcome measure.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Change from baseline in 15 minutes | -0.21 (0.101) | -0.10 (0.099)
  Change from baseline in 30 minutes | -0.22 (0.100) | -0.19 (0.099)
  Change from baseline in 60 minutes | -0.32 (0.104) | -0.32 (0.102)
  Change from baseline in 120 minutes | -0.47 (0.110) | -0.46 (0.108)
  Change from baseline in 180 minutes | -0.58 (0.126) | -0.57 (0.124)
  Change from baseline in 240 minutes | -0.64 (0.126) | -0.60 (0.124)

11. Secondary Outcome: Nasal Congestion Severity Assessment
Description: Participants self-assessed nasal congestion severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at baseline and at 15, 30, 60, 120,180 and 240 minutes post product administration. All nasal congestion severity assessment values were recorded in a questionnaire and tabulated. A reduction in severity score from baseline represented a better outcome measure.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Change from baseline in 15 minutes | -0.32 (0.086) | -0.31 (0.084)
  Change from baseline in 30 minutes | -0.59 (0.119) | -0.60 (0.115)
  Change from baseline in 60 minutes | -0.61 (0.127) | -0.68 (0.124)
  Change from baseline in 120 minutes | -0.91 (0.138) | -1.02 (0.134)
  Change from baseline in 180 minutes | -1.04 (0.156) | -1.14 (0.152)
  Change from baseline in 240 minutes | -1.19 (0.162) | -1.20 (0.157)

12. Secondary Outcome: Runny Nose Severity Assessment
Description: Participants self-assessed runny nose severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at baseline and at 15, 30, 60, 120,180 and 240 minutes post product administration. All runny nose severity assessment values were recorded in questionnaire and tabulated. A reduction in severity score from baseline represented a better outcome measure.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Change from baseline in 15 minutes | -0.20 (0.081) | -0.18 (0.080)
  Change from baseline in 30 minutes | -0.48 (0.116) | -0.32 (0.114)
  Change from baseline in 60 minutes | -0.54 (0.145) | -0.61 (0.143)
  Change from baseline in 120 minutes | -0.78 (0.148) | -0.65 (0.146)
  Change from baseline in 180 minutes | -0.89 (0.161) | -0.98 (0.159)
  Change from baseline in 240 minutes | -1.12 (0.149) | -0.97 (0.147)

13. Secondary Outcome: Sneezing Severity Assessment
Description: Participants self-assessed sneezing severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at baseline and at 15, 30, 60, 120,180 and 240 minutes post product administration. All sneezing severity assessment values were recorded in a questionnaire and tabulated. A reduction in severity score from baseline represented a better outcome measure.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Change from baseline in 15 minutes | -0.10 (0.089) | -0.24 (0.088)
  Change from baseline in 30 minutes | -0.25 (0.103) | -0.42 (0.102)
  Change from baseline in 60 minutes | -0.50 (0.126) | -0.80 (0.124)
  Change from baseline in 120 minutes | -0.67 (0.138) | -0.86 (0.136)
  Change from baseline in 180 minutes | -0.83 (0.138) | -1.03 (0.136)
  Change from baseline in 240 minutes | -0.88 (0.135) | -1.11 (0.133)

14. Secondary Outcome: Cough Severity Assessment
Description: Participants self-assessed cough severity using 4 points (0 = absent, 1 = mild, 2 = moderate, and 3 = severe) categorical scale at baseline and at 15, 30, 60, 120,180 and 240 minutes post product administration. All cough severity assessment values were recorded in a questionnaire and tabulated. A reduction in severity score from baseline represented a better outcome measure.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
Score on scale
  Change from baseline in 15 minutes | -0.11 (0.071) | -0.06 (0.078)
  Change from baseline in 30 minutes | -0.28 (0.077) | -0.25 (0.084)
  Change from baseline in 60 minutes | -0.49 (0.116) | -0.33 (0.126)
  Change from baseline in 120 minutes | -0.51 (0.109) | -0.45 (0.119)
  Change from baseline in 180 minutes | -0.53 (0.116) | -0.53 (0.127)
  Change from baseline in 240 minutes | -0.72 (0.131) | -0.59 (0.143)

15. Secondary Outcome: Body Temperature Reduction
Description: Summary statistics for body temperature was presented at baseline and at 15, 30, 60, 120,180 and 240 minutes post treatment. Wilcoxon Rank Sum test was used to investigate if there are any significant treatment differences.
Time Frame: Change from baseline in 15, 30, 60,120, 180, and 240 minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: °C (degree Celsius)
Arm/Group | Test Tablet | Placebo
Number analyzed (Participants) | 25 | 27
°C (degree Celsius)
  Change from baseline to 15 minutes | -0.02 (0.070) | 0.01 (0.047)
  Change from baseline to 30 minutes | -0.03 (0.080) | -0.01 (0.071)
  Change from baseline to 60 minutes | -0.04 (0.081) | 0.01 (0.049)
  Change from baseline to 120 minutes | -0.09 (0.079) | -0.04 (0.065)
  Change from baseline to 180 minutes | -0.14 (0.060) | -0.09 (0.067)
  Change from baseline to 240 minutes | -0.08 (0.058) | -0.11 (0.066)

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of the study until 5 days following last administration of the investigational product
Arm/Group | Test Tablet | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27
Other Adverse Events (participants affected / at risk) | 1/25 | 3/27
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Tablet (N=25) | Placebo (N=27)
GINGIVAL SWELLING (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.